CLINICAL TRIAL: NCT02379871
Title: The Effects of Mid-thoracic Manipulation on Heart Rate Variability.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mount St. Mary's College, Los Angeles, CA (Other)
Responsible Party: Principal Investigator, Derrick Sueki, Principal Investigator, Mount St. Mary's College, Los Angeles, CA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MountSMCLA 2
Record Dates: First submitted 2015-02-16; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Neurophysiological Mechanisms Underlying Spinal Manipulation
Keywords: Thoracic Spinal Manipulation, Autonomic Nervous System

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): While lying in supine, subjects will receive a single posterior to anterior directed spinal manipulation to the mid-thoracic region (T4-5).
  Interventions: Other: Experimental Group
- Sham Group (Sham Comparator): Sham group will procedures will be identical with the exception of the spinal manipulation intervention. Sham shall not receive the spinal manipulation intervention.
  Interventions: Other: Sham Group

INTERVENTIONS:
Other: Experimental Group — Supine mid-thoracic spinal manipulation to the T4/5 region
  Arms: Experimental Group
Other: Sham Group — Subject will be positioned in supine identical to the experimental group, but no spinal manipulation will be delivered.
  Arms: Sham Group

SUMMARY:
The topic of spinal manipulation (SM) has been a source of increasing research over the past decade. Research has focused primarily upon the functional and clinical outcomes associated with SM. The physiological mechanisms underlying the clinical changes experienced following SM are still largely unknown. Current thought suggests that SM may have an effect upon the neurophysiological system, specifically the autonomic nervous system. The purpose of this study will be to explore the effects of SM upon the autonomically regulated cardiovagal response.

DETAILED DESCRIPTION:
Subjects will be asked to report to the exercise room at Mount St. Mary's College in the physical therapy building for only one session lasting approximately 15-20 minutes. The subject will fill out a small questionnaire to rule out any health conditions, which would exclude them. The subject will next be informed about the methods and nature of the study after which they will be asked to sign an informed consent form. Once signed, the subject will be included into the study and will be randomized to either the manipulative group, the sham manipulation group or the control group. The Biocomm HRV Live! heart rate variability monitor will be attached to the subject's wrist who will then be asked to lie supine on a treatment table for five minutes. The monitor is composed of a simple recording electrode that is secured to the wrist with either tape or a band. At this time the principal investigator will perform a manual technique on the individuals randomized into the manipulation group. The subject will be asked to place his/her hands behind her neck with her elbows aligned with their body. The principal investigator will then slightly roll the subject's torso towards herself while placing her left hand in a flexed position underneath the subject's spine at the T4-T5 level. The principal investigator will then flex the subject's thoracic spine by placing her right forearm on the subject's elbows and asking the subject to do a slight crunch. Then the principal investigator will apply the high velocity-low amplitude thrust in the anterior-posterior direction through the subject's forearms and over her left hand under the subject. For the sham manipulation group, no force will be placed through the elbows, but all other aspects of positioning will be the same as the manipulation group. The control group will be asked to link their fingers behind their neck and rest for one minute. Following the intervention, the subject will be asked to lie quietly in supine for an additional ten minutes to record post manipulation responses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* History of back surgeries, osteopenia, osteoporosis, spinal fractures, rib fractures, chronic pain over three months, or heart conditions. Subjects will also be excluded if they are currently taking or have a significant history of taking steroid or anticoagulant medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) | 5 minutes pre-intervention (baseline), immediately post intervention, 10 minutes post intervention
  Change in heart rate variability via continuous heart rate monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Derrick Sueki, DPT, Principal Investigator — Mount St. Mary's College, Los Angeles, CA
Locations (1):
- Mount St. Mary's College, Los Angeles, California, United States